CLINICAL TRIAL: NCT01831765
Title: Efficacy and Safety of FIAsp Compared to Insulin Aspart Both in Combination With Insulin Detemir in Adults With Type 1 Diabetes
Acronym: onset® 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-3852; 2010-024049-53 (EudraCT Number); U1111-1118-2442 (Other: WHO)
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Meal time FIAsp and insulin detemir (Experimental)
  Interventions: Drug: Faster-acting insulin aspart; Drug: insulin detemir
- Meal time insulin aspart and insulin detemir (Active Comparator)
  Interventions: Drug: insulin detemir; Drug: insulin aspart
- Post meal FIAsp and insulin detemir (Experimental)
  Interventions: Drug: insulin detemir; Drug: Faster-acting insulin aspart

INTERVENTIONS:
Drug: Faster-acting insulin aspart — Injected subcutaneously (s.c., under the skin), dose individually adjusted. Meal time dosing is defined as injecting 0-2 minutes before the meal.
  Arms: Meal time FIAsp and insulin detemir
Drug: insulin detemir — Injected subcutaneously (s.c., under the skin), dose individually adjusted. Administrated once or twice daily.
Drug: insulin aspart — Injected subcutaneously (s.c., under the skin), dose individually adjusted.
  Arms: Meal time insulin aspart and insulin detemir
Drug: Faster-acting insulin aspart — Injected subcutaneously (s.c., under the skin), dose individually adjusted. Post meal time dosing is defined as injecting 20 minutes after the start of the meal.
  Arms: Post meal FIAsp and insulin detemir

SUMMARY:
This trial is conducted in Europe and the United States of America (USA). The aim of the trial is to investigate efficacy and safety of FIAsp (faster-acting insulin aspart) compared to insulin aspart, both in combination with insulin detemir in adults with type 1 diabetes. This trial consists of two periods: a 26 week treatment period followed by a 26 week additional treatment period.

ELIGIBILITY:
Inclusion Criteria: - Type 1 diabetes (diagnosed clinically) for 12 months or longer at the time of screening (Visit 1) - Currently treated with a basal-bolus insulin regimen for at least 12 months prior to screening (Visit 1) - Currently treated with a basal insulin analogue (any regimen of insulin detemir or insulin glargine) for at least 4 months prior to screening (Visit 1) - HbA1c 7.0-9.5% (53-80 mmol/mol) (both inclusive) as assessed by central laboratory - Body Mass Index (BMI) below or equal to 35.0 kg/m^2 Exclusion Criteria: - Use of any anti-diabetic drug other than insulin within the last 3 months prior to screening (Visit 1) - Recurrent severe hypoglycaemia (more than one severe hypoglycaemic event during the last 12 months) or hypoglycaemic unawareness as judged by the Investigator, or hospitalisation for diabetic ketoacidosis during the previous 6 months prior to screening (Visit 1) - Cardiovascular disease, within the last 6 months prior to screening (Visit 1), defined as stroke, decompensated heart failure New York Heart Association (NYHA) class III or IV, myocardial infarction, unstable angina pectoris, coronary arterial bypass graft or angioplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1290 (Actual)
Dates: Start 2013-08-26 (Actual); Primary Completion 2015-05-12 (Actual); Study Completion 2015-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (157):
- United States (90):
  - Novo Nordisk Investigational Site, Mobile, Alabama
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Fullerton, California
  - Novo Nordisk Investigational Site, Inglewood, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, La Mesa, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, North Hollywood, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, Poway, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Santa Barbara, California
  - Novo Nordisk Investigational Site, Ventura, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Newark, Delaware
  - Novo Nordisk Investigational Site, Boca Raton, Florida
  - Novo Nordisk Investigational Site, Coral Gables, Florida
  - Novo Nordisk Investigational Site, Fleming Island, Florida
  - Novo Nordisk Investigational Site, Fort Lauderdale, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Sanford, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Dunwoody, Georgia
  - Novo Nordisk Investigational Site, Lawrenceville, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Nampa, Idaho
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Crystal Lake, Illinois
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, Muncie, Indiana
  - Novo Nordisk Investigational Site, Lenexa, Kansas
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Portland, Maine
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Waltham, Massachusetts
  - Novo Nordisk Investigational Site, Worcester, Massachusetts
  - Novo Nordisk Investigational Site, Kalamazoo, Michigan
  - Novo Nordisk Investigational Site, Eagan, Minnesota
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, Springfield, Missouri
  - Novo Nordisk Investigational Site, Butte, Montana
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Henderson, Nevada
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Hoboken, New Jersey
  - Novo Nordisk Investigational Site, Jersey City, New Jersey
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Rochester, New York
  - Novo Nordisk Investigational Site, Smithtown, New York
  - Novo Nordisk Investigational Site, Staten Island, New York
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Morehead City, North Carolina
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Mentor, Ohio
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Jenkintown, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Greenville, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Amarillo, Texas
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Beaumont, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Lubbock, Texas
  - Novo Nordisk Investigational Site, Plano, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Magna, Utah
  - Novo Nordisk Investigational Site, Olympia, Washington
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Spokane, Washington
- Belgium (5):
  - Novo Nordisk Investigational Site, Bonheiden
  - Novo Nordisk Investigational Site, Brussels
  - Novo Nordisk Investigational Site, Edegem
  - Novo Nordisk Investigational Site, Ghent
  - Novo Nordisk Investigational Site, Leuven
- Canada (10):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Victoria, British Columbia
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Mississauga, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Montreal, Quebec
  - Novo Nordisk Investigational Site, Sherbrooke, Quebec
  - Novo Nordisk Investigational Site, Québec
- Czechia (3):
  - Novo Nordisk Investigational Site, Brno
  - Novo Nordisk Investigational Site, Hradec Králové
  - Novo Nordisk Investigational Site, Prague
- Finland (6):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Kerava
  - Novo Nordisk Investigational Site, Lappeenranta
  - Novo Nordisk Investigational Site, Raisio
  - Novo Nordisk Investigational Site, Tampere
  - Novo Nordisk Investigational Site, Turku
- Germany (23):
  - Novo Nordisk Investigational Site, Bad Mergentheim
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Damme
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Elsterwerda
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Fulda
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Lingen
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Neuwied
  - Novo Nordisk Investigational Site, Oldenburg
  - Novo Nordisk Investigational Site, Rehburg-Loccum
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Rostock
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
  - Novo Nordisk Investigational Site, Schweinfurt
  - Novo Nordisk Investigational Site, Völklingen
  - Novo Nordisk Investigational Site, Wangen
  - Novo Nordisk Investigational Site, Zwenkau
- Hungary (5):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
  - Novo Nordisk Investigational Site, Kaposvár
  - Novo Nordisk Investigational Site, Szeged
  - Novo Nordisk Investigational Site, Szombathely
- Poland (6):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Szczecin
  - Novo Nordisk Investigational Site, Warsaw
- United Kingdom (9):
  - Novo Nordisk Investigational Site, Bath
  - Novo Nordisk Investigational Site, Gillingham
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Guildford
  - Novo Nordisk Investigational Site, Inverness
  - Novo Nordisk Investigational Site, Ipswich
  - Novo Nordisk Investigational Site, Nottingham
  - Novo Nordisk Investigational Site, Portsmouth
  - Novo Nordisk Investigational Site, Sheffield

REFERENCES:
- [Background] Rose L, Kadowaki T, Pieber TR, Buchholtz K, Ekelund M, Gorst-Rasmussen A, Philis-Tsimikas A. Efficacy and Safety of Fast-Acting Insulin Aspart in People with Type 1 Diabetes Using Carbohydrate Counting: A Post Hoc Analysis of Two Randomised Controlled Trials. Diabetes Ther. 2019 Jun;10(3):1029-1041. doi: 10.1007/s13300-019-0608-4. Epub 2019 Apr 4. PMID 30949906
- [Result] Russell-Jones D, Bode BW, De Block C, Franek E, Heller SR, Mathieu C, Philis-Tsimikas A, Rose L, Woo VC, Osterskov AB, Graungaard T, Bergenstal RM. Fast-Acting Insulin Aspart Improves Glycemic Control in Basal-Bolus Treatment for Type 1 Diabetes: Results of a 26-Week Multicenter, Active-Controlled, Treat-to-Target, Randomized, Parallel-Group Trial (onset 1). Diabetes Care. 2017 Jul;40(7):943-950. doi: 10.2337/dc16-1771. Epub 2017 Mar 29. PMID 28356319
- [Result] Mathieu C, Bode BW, Franek E, Philis-Tsimikas A, Rose L, Graungaard T, Birk Osterskov A, Russell-Jones D. Efficacy and safety of fast-acting insulin aspart in comparison with insulin aspart in type 1 diabetes (onset 1): A 52-week, randomized, treat-to-target, phase III trial. Diabetes Obes Metab. 2018 May;20(5):1148-1155. doi: 10.1111/dom.13205. Epub 2018 Feb 4. PMID 29316130
- [Result] Bode BW, Bowering K, Russell-Jones D. Response to Comment on Russell-Jones et al. Diabetes Care 2017;40:943-950. Comment on Bowering et al. Diabetes Care 2017;40:951-957. Diabetes Care. 2018 Mar;41(3):e29-e30. doi: 10.2337/dci17-0051. No abstract available. PMID 29463670
- [Result] Haahr H, Pieber TR, Mathieu C, Gondolf T, Shiramoto M, Erichsen L, Heise T. Clinical Pharmacology of Fast-Acting Insulin Aspart Versus Insulin Aspart Measured as Free or Total Insulin Aspart and the Relation to Anti-Insulin Aspart Antibody Levels in Subjects with Type 1 Diabetes Mellitus. Clin Pharmacokinet. 2019 May;58(5):639-649. doi: 10.1007/s40262-018-0718-6. PMID 30402720
- [Result] Bowering K, Rodbard HW, Russell-Jones D, Bode B, Harris S, Piletic M, Heller S, Woo V, Babu V, Dethlefsen C, Mathieu C. Investigating the Association Between Baseline Characteristics (HbA1c and Body Mass Index) and Clinical Outcomes of Fast-Acting Insulin Aspart in People with Diabetes: A Post Hoc Analysis. Diabetes Ther. 2019 Feb;10(1):177-188. doi: 10.1007/s13300-018-0553-7. Epub 2018 Dec 13. PMID 30547388
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 281 sites, selected for recruitment, 165 sites in 9 countries enrolled subjects in the run-in period, of which 163 sites later assigned subjects to randomised treatment: Belgium:5 sites, Canada:12 sites, Czech Republic:5 sites; Finland:6 sites; Germany:25 sites; Hungary:5 sites; Poland:6 sites; United Kingdom:9 sites; United States:92 sites.
Pre-assignment Details: Eligible subjects received once/twice daily insulin detemir and NovoRapid®/NovoLog® during 8 week run-in period. In total, 1290 subjects entered the run-in period, of those147 subjects were run-in failures. Hence 1143 subjects entered the 26-week treatment period followed by a 26 week additional treatment period.
Groups:
- Faster Aspart (Meal): The subjects in this arm were administered mealtime faster aspart (100 U/mL) in combination with once or twice daily insulin detemir (100 U/mL) in a basal-bolus regimen for an initial 26 weeks treatment period + a 26-week additional treatment period. Mealtime faster aspart was administered subcutaneously (s.c., under the skin) 0-2 minutes before each main meal. Subjects who, prior to screening, had used the principles of flexible dosing based on the meal carbohydrate content, and who were assessed by the investigator to be adequately trained in this method, were to continue using this method for bolus adjustment during the treatment period. All other subjects were to use a predefined bolus dosing algorithm to adjust the bolus dose during the treatment period. Additional bolus dosing was allowed at the investigator's recommendation.
- Faster Aspart (Post): The subjects in this arm were administered postmeal faster aspart (100 U/mL) in combination with once or twice daily insulin detemir (100 U/mL) in a basal-bolus regimen for an initial 26 weeks treatment period. Postmeal faster aspart was administered subcutaneously (s.c., under the skin) 20 minutes after the start of the meal. Subjects who, prior to screening, had used the principles of flexible dosing based on the meal carbohydrate content, and who were assessed by the investigator to be adequately trained in this method, were to continue using this method for bolus adjustment during the treatment period. All other subjects were to use a predefined bolus dosing algorithm to adjust the bolus dose during the treatment period. Additional bolus dosing was allowed at the investigator's recommendation.
- NovoRapid (Meal): The subjects in this arm were administered mealtime NovoRapid®/NovoLog®, 100 U/mL in combination with once or twice daily insulin detemir (100 U/mL) in a basal-bolus regimen for an initial 26 weeks treatment period + a 26-week additional treatment period. Mealtime NovoRapid®/NovoLog® was administered subcutaneously (s.c., under the skin) 0-2 minutes before each main meal. Subjects who, prior to screening, had used the principles of flexible dosing based on the meal carbohydrate content, and who were assessed by the investigator to be adequately trained in this method, were to continue using this method for bolus adjustment during the treatment period. All other subjects were to use a predefined bolus dosing algorithm to adjust the bolus dose during the treatment period. Additional bolus dosing was allowed at the investigator's recommendation.
Period: Overall Study
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Started | 381 | 382 | 380
Completed 26 Weeks | 351 | 355 | 356
Completed 52 Weeks | 337 | 0 (This arm did not continue in the trial after 26 weeks ( 26 to 52 weeks).) | 338
Completed | 337 | 355 | 338
Not Completed | 44 | 27 | 42
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Other, sponsor withdrew subject | 0 | 1 | 0
Not completed — Pregnancy | 1 | 1 | 2
Not completed — Death | 0 | 1 | 1
Not completed — Other, site closed | 1 | 1 | 0
Not completed — Adverse Event | 5 | 3 | 3
Not completed — Withdrawal by Subject | 22 | 7 | 17
Not completed — Withdrawal criteria | 12 | 10 | 16
Not completed — Lost to Follow-up | 2 | 3 | 3

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomised subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal) | Total
Number analyzed (Participants) | 381 | 382 | 380 | 1143
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.1 (13.8) | 43.5 (13.7) | 43.7 (14) | 44.4 (13.9)
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 346 | 359 | 352 | 1057
  From 65-85 years | 35 | 23 | 28 | 86
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 163 | 142 | 471
  Male | 215 | 219 | 238 | 672
Body Weight [Mean (Standard Deviation); unit: Kg] | 78.56 (14.89) | 80.49 (15.93) | 80.15 (15.21) | 79.73 (15.36)
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin] | 7.62 (0.71) | 7.63 (0.72) | 7.58 (0.68) | 7.61 (0.70)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Glycosylated Haemoglobin)
Description: Change from baseline in HbA1c after 26 weeks of randomised treatment.
Time Frame: Week 0, week 26
Population: The FAS included all randomised subjects. For this endpoint, baseline and week 26 have been presented, where week 26 data is end of trial containing last available measurement.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 381 | 382 | 380
Percentage of glycosylated haemoglobin
  Week 0 (Baseline) | 7.62 (0.71) | 7.63 (0.72) | 7.58 (0.68)
  Week 26 | 7.31 (0.77) | 7.51 (0.77) | 7.42 (0.78)
Statistical Analysis 1: Comparison: Faster Aspart (Meal) vs NovoRapid (Meal); Change from baseline in HbA1c analysed using a mixed effect model for repeated measurements including visit 14, 18, 22, 26, 30, 34 and 36. The model included treatment, region and strata (combination of bolus adjusting method, basal treatment regimen and continuous glucose monitoring (CGM) and frequently sampled meal test subgroup) as fixed effects, subject as random effect, baseline HbA1c as covariate and interaction between all fixed effects and visit, and between the covariate and visit; Test type: Non-Inferiority or Equivalence — The assessment was done by comparing the difference of faster aspart vs. NovoRapid®/NovoLog® in change from baseline in HbA1c after 26 weeks of randomised treatment to a non-inferiority limit of 0.4%; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.23 to -0.07]
Statistical Analysis 2: Comparison: Faster Aspart (Post) vs NovoRapid (Meal); Change from baseline in HbA1c analysed using a mixedeffect model for repeated measurements including visit 14, 18, 22, 26, 30, 34 and 36. The model included treatment, region and strata (combination of bolus adjusting method, basal treatment regimen and continuous glucose monitoring (CGM) and frequently sampled meal test subgroup) as fixed effects, subject as random effect, baseline HbA1c as covariate and interaction between all fixed effects and visit, and between the covariate and visit; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.04 to 0.12]

2. Secondary Outcome: Change From Baseline in 2-hour PPG (Postprandial Glucose) Increment (Meal Test)
Description: Change from baseline in 2-hour PPG increments after 26 weeks of randomised treatment (meal test).
Time Frame: Week 0, week 26
Population: The FAS included all randomised subjects. For this endpoint, baseline and week 26 have been presented, where week 26 data is end of trial containing last available measurement. At baseline (week 0) 379, 377, 375 and 381, 382, 380 subjects at week 26 were analysed for faster aspart (meal), faster aspart (post) and Novorapid (meal) arms respectively.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 381 | 382 | 380
mmol/L
  Week 0: Baseline: number analyzed (Participants) | 379 | 377 | 375
  Week 0: Baseline | 6.06 (5.16) | 6.06 (4.9) | 6.24 (4.81)
  Week 26 | 5.88 (4.67) | 6.73 (4.67) | 6.55 (4.78)

3. Secondary Outcome: Change From Baseline in HbA1c (Post Meal Arm)
Description: Change from baseline in HbA1c (post meal arm) after 26 weeks of randomised treatment.
Time Frame: Week 0, week 26
Population: This endpoint was summarised using the FAS, which included all randomised subjects. For this endpoint, baseline and week 26 have been presented, where week 26 data is end of trial containing last available measurement.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin
Arm/Group | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 382 | 380
Percentage of glycosylated haemoglobin
  Week 0 (baseline) | 7.63 (0.72) | 7.58 (0.68)
  Week 26 | 7.51 (0.77) | 7.42 (0.78)

4. Secondary Outcome: Number of Treatment Emergent Confirmed Hypoglycaemic Episodes
Description: Observed rate of treatment emergent severe or BG confirmed hypoglycaemic events per 100 patient years of exposure (PYE) from baseline until week 26. A hypoglycaemic episode was defined as treatment emergent if the onset of the episode was on or after the first day of exposure to randomised treatment and no later than 1 day after the last day of randomised treatment. Severe or BG confirmed is an episode that is severe according to the American Diabetes Association (ADA) classification (an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or BG confirmed by a PG value <3.1 mmol/L (56 mg/dL) with or without symptoms consistent with hypoglycaemia.
Time Frame: From baseline until week 26
Population: The safety analysis set included all subjects receiving at least one dose of trial product/its comparator and contributed to the evaluation "as treated". Five (5) subjects randomised to the faster aspart (post) group have consistently taken their bolus insulin before meals throughout the trial and are handled as treated with faster aspart (meal).
Measure: Number; unit: event rate/100 patient yrs of exposure
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 386 | 377 | 380
event rate/100 patient yrs of exposure | 5899 | 5443 | 5865

5. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight after 26 weeks of randomised treatment.
Time Frame: Week 0, week 26
Population: The FAS included all randomised subjects. For this endpoint baseline, and week 26 have been presented, where week 26 data is end of trial containing last available measurement. At baseline (week 0) 381, 382, 378 and 381, 382, 380 subjects at week 26 were analysed for faster aspart (meal), faster aspart (post) and Novorapid (meal) arms respectively.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 381 | 382 | 380
Kg
  Week 0: Baseline | 78.56 (14.89) | 80.49 (15.93) | 80.15 (15.21)
  Week 26 | 79.21 (15.25) | 81.17 (16.45) | 80.69 (15.44)

6. Secondary Outcome: Frequency of Adverse Events
Description: All treatment emergent adverse events (TEAEs) from baseline until 52 weeks of randomised treatment. A TEAE was defined as an event that had an onset date on or after the first day of exposure to randomised treatment, and no later than 7 days after the last day of randomised treatment.
Time Frame: After 52 weeks of randomised treatment
Population: as for outcome 4
Measure: Number; unit: event /100 patient yrs of exposure
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 386 | 377 | 380
event /100 patient yrs of exposure | 445.8 | 441 | 411

7. Secondary Outcome: Change in HbA1c
Description: Change from baseline in HbA1c (%) after 52 weeks of randomised treatment.
Time Frame: Week 0, week 52
Population: The FAS included all randomised subjects. The statistical evaluation of the FAS was to follow the ITT principle and subjects contributed to the evaluation 'as randomised'. For this endpoint, baseline and week 52 have been presented, where week 52 data is the end of trial containing last available measurement.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin
Arm/Group | Faster Aspart (Meal) | NovoRapid (Meal)
Number analyzed (Participants) | 381 | 380
Percentage of glycosylated haemoglobin
  Week 0 (baseline) | 7.62 (0.71) | 7.58 (0.68)
  Week 52 | 7.51 (0.83) | 7.58 (0.86)

8. Secondary Outcome: Change in PPG (Postprandial Glucose)
Description: Change from baseline in PPG and PPG increment (meal test) after 52 weeks of randomised treatment.
Time Frame: Week 0, week 52
Population: The FAS included all randomised subjects. The number of subjects with data available for PPG at 120 mins at baseline were 379, 379 and 380, 380 at week 52 and for PPG increment (120 mins) at baseline were 379, 375 and 381, 380 at week 26 for faster aspart (meal) and Novorapid (meal) respectively.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | NovoRapid (Meal)
Number analyzed (Participants) | 381 | 380
mmol/L
  PPG at 120 minutes (Baseline): number analyzed (Participants) | 379 | 379
  PPG at 120 minutes (Baseline) | 14.51 (6.09) | 14.14 (5.69)
  PPG at 120 minutes (Week 52): number analyzed (Participants) | 380 | 380
  PPG at 120 minutes (Week 52) | 14.26 (5.76) | 14.51 (6.02)
  PPG increment at 120 mins (Baseline): number analyzed (Participants) | 379 | 375
  PPG increment at 120 mins (Baseline) | 6.06 (5.16) | 6.24 (4.81)
  PPG increment at 120 mins(Week 52) | 5.71 (4.92) | 6.14 (4.86)

ADVERSE EVENTS:
Time Frame: Until 52 weeks (26+26) weeks of treatment + 7 days followup for faster aspart (meal) and NovoRapid®(meal) or until 26 weeks of treatment + 7 days followup for faster aspart (post) + 30 day follow-up period for cardio-vascular related events.
Description: The safety analysis set included all subjects receiving at least one dose of trial product/ its comparator and contributed to the evaluation "as treated". A TEAE was defined as an event recorded from the first day of exposure to trial product and no later than post-treatment follow-up visit (7 days). Five (5) subjects randomised to the faster aspart (post) group have consistently taken their bolus insulin before meals throughout the trial and are handled as treated with faster aspart (meal).
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Serious Adverse Events (participants affected / at risk) | 35/386 | 28/377 | 33/380
Other Adverse Events (participants affected / at risk) | 252/386 | 189/377 | 236/380
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faster Aspart (Meal) (N=386) | Faster Aspart (Post) (N=377) | NovoRapid (Meal) (N=380)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiovascular evaluation (Investigations) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Coronary revascularisation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 12 (16) | 11 (11) | 10 (10)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 5 (8) | 3 (3) | 4 (5)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peritoneal fibrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wrong drug administered (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faster Aspart (Meal) (N=386) | Faster Aspart (Post) (N=377) | NovoRapid (Meal) (N=380)
Back pain (Musculoskeletal and connective tissue disorders) | 28 (36) | 15 (17) | 20 (22)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 12 (13) | 20 (21)
Diarrhoea (Gastrointestinal disorders) | 27 (34) | 11 (11) | 27 (33)
Gastroenteritis (Infections and infestations) | 20 (25) | 8 (8) | 17 (21)
Headache (Nervous system disorders) | 37 (70) | 26 (41) | 45 (79)
Influenza (Infections and infestations) | 22 (30) | 11 (12) | 37 (54)
Nasopharyngitis (Infections and infestations) | 128 (214) | 90 (111) | 120 (174)
Nausea (Gastrointestinal disorders) | 28 (36) | 18 (29) | 23 (34)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17 (22) | 16 (21) | 23 (30)
Sinusitis (Infections and infestations) | 19 (21) | 7 (7) | 28 (37)
Upper respiratory tract infection (Infections and infestations) | 56 (75) | 28 (31) | 40 (61)
Urinary tract infection (Infections and infestations) | 20 (25) | 15 (20) | 18 (29)
Vomiting (Gastrointestinal disorders) | 19 (23) | 15 (16) | 25 (30)
Wrong drug administered (Injury, poisoning and procedural complications) | 22 (31) | 18 (20) | 23 (28)

LIMITATIONS AND CAVEATS:
Limitations of the trial such as small numbers of subjects analysed or technical problems leading to unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more manuscripts for publication will be prepared collaboratively between Investigator(s) and Novo Nordisk.

Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property.